CLINICAL TRIAL: NCT00992394
Title: Randomized Open-label Study Comparing 2 Different Strategies For Management Of Subjects With Plaque Psoriasis Who Have Responded To Etanercept Treatment
Brief Title: Study Comparing 2 Different Strategies For Management of Subjects With Plaque Psoriasis Who Have Responded to Etanercept
Acronym: ReSPONSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881X1-4535; B1801021 (Other: Alias Study Number); 2008-004439-39 (EudraCT Number)
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis
Keywords: Plaque psoriasis - etanercept - response maintenance
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other): Subjects randomized to arm 1 stop their etanercept treatment on entry into the study and may be retreated by etanercept 50 mg once weekly after medical review and agreement between the subject and the investigator
  Interventions: Drug: etanercept
- Arm 2 (Other): Subjects randomized to arm 2 in which subjects continue on treatment with etanercept at 25 mg once weekly, but with the option to have their drug treatment increased to 50 mg once weekly after medical review and agreement between the subject and the investigator
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — etanercept 50 mg once weekly as requested.
  Arms: Arm 1
Drug: etanercept — etanercept 25 mg or 50 mg as requested.
  Arms: Arm 2

SUMMARY:
This study proposes to compare 2 different methods for managing a subject with psoriasis who has achieved good disease control, as defined by a clinical response with a Physician Global Assessment (PGA) inferior or equal to 1 at the screening visit, on etanercept treatment.

The first method involves stopping etanercept treatment on entry into the study, with the option to reinitiate etanercept at 50 mg once weekly after medical review and agreement between the subject and the investigator. The second method involves continuing on etanercept at 25 mg once weekly, with the option to increase the dose to 50 mg once weekly after medical review and agreement between the subject and the investigator. Subjects will be randomized into one of these two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) years of age or older at the time of consent.
* Previously treated with etanercept for chronic plaque psoriasis for at least 12 weeks prior to the screening visit and received a total weekly dose of 50 mg per week for at least the 6 weeks preceding the day of the screening visit
* Having shown clinical response with a PGA inferior or equal to 1 at the screening visit.
* PGA inferior or equal to 1 at the baseline visit.

Exclusion Criteria:

* Evidence of skin conditions (eg, eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Evidence of active or previously known medical history of inflammatory arthritis (eg, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis).
* Any biologics other than etanercept within the 20 weeks prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- France (10):
  - Centre Hopitalier St Jacques (Place St Jacques), Besançon
  - CHU Dupuytren, Limoges
  - Service de Chirurgie Infantile, Lyon
  - C.H.U Nantes, Nantes
  - CHU de l Archet, Nice
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - C.H.U de Reims, Reims
  - Hôpital Purpan, Toulouse
- Germany (7):
  - Klinik fuer Dermatologie, Allergologie und Venerologie, Berlin
  - St. Josef-Klinikum, Bochum
  - Universitaetsklinikum Erlangen Hautklinik im Internistischen Zentrum, Erlangen
  - J. W. Goethe Universitaet Frankfurt, Zentrum fuer Dermatologie und Venerologie, Frankfurt am Main
  - Klinikum der Albert-Ludwigs-Universitaet, Freiburg im Breisgau
  - Universitätsklinikum-Eppendorf Martinistr. 20, Hamburg 20158, Hamburg
  - Dermatologische Gemeinschaftspraxis Rosenbach, Osnabrück
- Greece (2):
  - "Andreas Sygros" Hospital, Athens
  - Papageorgiou General Peripheral Hospital of Thessaloniki, Thessaloniki
- Hungary (4):
  - Semmelweis Egyetem, Bor-, Nemikortani es Boronkologiai Klinika, Budapest
  - Debreceni Egyetem Orvos-és Egészségtudományi Centrum, Debrecen
  - Miskolci Egeszsegugyi Kozpont, Miskolc
  - SZTE, Szent-Gyorgyi Albert Klinikai Kozpont, Borgyogyaszati es Allergologiai Klinika, Szeged
- Italy (3):
  - Clinica Dermatologica - Universita' di Catania, Catania
  - Centro di Ricerca Clinica Fondazione Universita' degli Studi Gabriele D'Annunzio, Chieti
  - U.O. Dermatologia, Parma
- Spain (6):
  - Hospital General Universitario Alicante C/ Maestro Alonso, 1, Alicante, Alicante
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Fundacion Hospital Alcorcon, Alcorcón, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Virgen de la VICTORIA, Málaga, Malaga
- Turkey (Türkiye) (11):
  - Istanbul Universitesi, Istanbul, Capa
  - Gulhane Askeri Tip Akademisi Tip Fakultesi, Ankara, Etlik
  - Gulhane Askeri Tip Fakultesi, Ankara, Etlik
  - Gulhane Military Medical Academy, Faculty of Medicine, Ankara, Etlik
  - Bezm-i Alem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul, Fatih
  - Uludag Universitesi, Bursa, Gorukle
  - T.C. Saglik Bakanligi Marmara Universitesi Egitim ve Arastirma Hastanesi Dermatoloji Anabilim Dali, Pendik, Istanbul
  - Gazi Universitesi, Ankara, Sihhiye
  - Hacettepe Universitesi, Ankara, Sihhiye
  - Hacettepe Universitesi, Ankara
  - Ege Universitesi Tip Fakultesi Dermatoloji Anabilim Dali, Bornova / Izmir
- Sheikh Khalifa Medical City, Abu Dhabi, UAE, United Arab Emirates
- United Kingdom (2):
  - Harrogate District Hospital, Harrogate, Harrogate
  - Whipps Cross Hospital, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881X1-4535&StudyName=Study%20Comparing%202%20Different%20Strategies%20For%20Management%20of%20Subjects%20With%20Plaque%20Psoriasis%20Who%20Have%20Responded%20to%20Etanercept

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter open label, randomized study screened 209 participants in 44 sites.
Pre-assignment Details: Psoriasis participants who had responded to initial treatment with ETN were enrolled in this study. Participants were randomized to 2 groups: Stop arm, stopped etanercept (ETN) treatment on study entry and could be retreated with ETN 50 mg once weekly. Maintenance arm, continued ETN treatment at 25 mg once weekly, but could increase dose to 50 mg.
Groups:
- Stop Arm: Participants randomized to stop their etanercept treatment on entry into the study and could be retreated by etanercept 50 mg once weekly after medical review and agreement between the participant and the investigator
- Maintenance Arm: Participants randomized to continue on treatment with etanercept at 25 mg once weekly, but with the option to have their drug treatment increased to 50 mg once weekly after medical review and agreement between the participant and the investigator
Period: Overall Study
Arm/Group | Stop Arm | Maintenance Arm
Started | 88 | 86
Safety Population | 87 | 84
mITT Population | 86 | 84
Completed | 64 | 72
Not Completed | 24 | 14
Not completed — Lack of Efficacy | 6 | 3
Not completed — Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 2 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other event | 1 | 0

BASELINE CHARACTERISTICS:
Population: A total of 174 subjects were randomized.Three subjects were randomized but did not take at least 1 dose of investigational product, and were therefore excluded from the safety population. One subject was excluded from the mITT population. The reason for exclusion was lack of at least one post-baseline PGA.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stop Arm | Maintenance Arm | Total
Number analyzed (Participants) | 87 | 84 | 171
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.39 (14.10) | 47.71 (13.77) | 49.08 (13.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 58 | 53 | 111

OUTCOME MEASURES:

1. Primary Outcome: Time-Normalized Area Under Curve (AUC) of Physician Global Assessment (PGA) of Psoriasis Score at Week 52
Description: PGA psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration and scaling across all psoriatic lesions. PGA of Psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). 'Clear' and "Almost clear' includes all participants who were scored as a 0 or 1. For participants who discontinued the study before week 52, the final PGA score was carried forward to the remaining time points before calculating the 52-week AUC. The AUC was calculated on the PGA score profile with the method of trapeziums from baseline visit to visit 52. The time-normalized AUC is defined as the ratio between AUC and the expected treatment period (days): AUC/ 52 weeks*7days + 1.
Time Frame: Week 52
Population: The modified intent-to-treat (mITT) population was the primary efficacy population and corresponded to all randomized subjects who had a baseline PGA and at least one postbaseline PGA. Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Units on a scale | 1.64 (0.75) | 1.33 (0.76)

2. Secondary Outcome: Time-Normalized Area Under Curve (AUC) of Dermatology Life Quality Index (DLQI) at Week 52
Description: DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
Time Frame: Week 52
Population: The modified intent-to-treat (mITT) population was the primary efficacy population and corresponded to all randomized subjects who had a baseline PGA and at least one postbaseline PGA.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Units on a scale | 4.07 (4.21) | 2.96 (3.23)

3. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): The Overall Appearance of Skin, at Baseline, Before Retreatment, and at the End of Retreatment
Description: Participants completed a satisfaction survey at baseline and throughout the study. Participants were asked to rate, based on their experience during the past week, how satisfied or dissatisfied they were with their psoriasis therapy in general. Responses were based on a 5-point scale: Very dissatisfied (0) to very satisfied (4), and never had this problem (5).
Time Frame: Baseline to Week 52
Population: mITT population was the primary efficacy population and corresponded to all randomized subjects who had a baseline PGA and at least one postbaseline PGA.
Measure: Number; unit: Number of participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of participants
  Baseline, Subjects Satisfied | 66 | 67
  Prior to Re-treatment, Cycle 1 | 15 | 5
  End of Re-treatment, Cycle 1 | 31 | 12
  Prior to Re-treatment, Cycle 2 | 5 | 1
  End of re-treatment, Cycle 2 | 10 | 2

4. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Flaking Skin, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 60 | 59
  Prior to Re-treatment, Cycle 1, Satisfied | 12 | 4
  End of Re-treatment, Cycle 1, satisfied | 26 | 11
  Prior to Re-treatment, Cycle, 2, Satisfied | 5 | 1
  End of Re-treatment, Cycle 2, Satisfied | 8 | 2

5. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Redness of the Skin, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 62 | 59
  Prior to Re-treatment, Cycle 1, Satisfied | 14 | 4
  End of Re-treatment, Cycle 1, Satisfied | 27 | 10
  Prior to Re-treatment, Cycle 2, Satisfied | 4 | 1
  End of Re-treatment, Cycle 2, Satisfied | 8 | 2

6. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Tightness of the Skin, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 61 | 54
  Prior to Re-treatment, Cycle 1, Satisfied | 17 | 5
  End of Re-treatment, Cycle 1, Satisfied | 30 | 9
  Prior to Re-treatment, Cycle 2, Satisfied | 6 | 2
  End of Re-treatment, Cycle 2, Satisfied | 10 | 0

7. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Bleeding of the Skin, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 45 | 37
  Prior to Re-treatment, Cycle 1, Satisfied | 17 | 11
  End of Re-treatment, Cycle 1, Satisfied | 22 | 10
  Prior to Re-treatment, Cycle 2, Satisfied | 7 | 2
  End of Re-treatment, Cycle 2, Satisfied | 10 | 2

8. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Burning Sensation in the Skin, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 51 | 39
  Prior to Re-treatment, Cycle 1, Satisfied | 14 | 6
  End of Re-treatment, Cycle 1, Satisfied | 23 | 8
  Prior to Re-treatment, Cycle 2, Satisfied | 4 | 1
  End of Re-treatment, Cycle 2, Satisfied | 10 | 2

9. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Skin Pain, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 47 | 44
  Prior to Re-treatment, Cycle 1, Satisfied | 13 | 7
  End of Re-treatment, Cycle 1, Satisfied | 24 | 8
  Prior to Re-treatment, Cycle 2, Satisfied | 5 | 1
  End of Re-treatment, Cycle 2, Satisfied | 9 | 1

10. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Joint Pain, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 33 | 23
  Prior to Re-treatment, Cycle 1, Satisfied | 7 | 7
  End of Re-treatment, Cycle 1, Satisfied | 14 | 7
  Prior to Re-treatment, Cycle 2, Satisfied | 5 | 2
  End of Re-treatment, Cycle 2, Satisfied | 7 | 1

11. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Your Comfort Level With Your Personal Appearance, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 64 | 58
  Prior to Re-treatment, Cycle 1, Satisfied | 17 | 6
  End of Re-treatment, Cycle 1, Satisfied | 35 | 8
  Prior to Re-treatment, Cycle 2, Satisfied | 8 | 1
  End of Re-treatment, Cycle 2, Satisfied | 10 | 2

12. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Anxiety, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 43 | 36
  Prior to Re-treatment, Cycle 1, Satisfied | 13 | 6
  End of Re-treatment, Cycle 1, Satisfied | 17 | 5
  Prior to Re-treatment, Cycle 2, Satisfied | 5 | 2
  End of Re-treatment, Cycle 2, Satisfied | 5 | 1

13. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Depression, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 39 | 31
  Prior to Re-treatment, Cycle 1, Satisfied | 15 | 5
  End of Re-treatment, Cycle 1, Satisfied | 17 | 3
  Prior to Re-treatment, Cycle 2, Satisfied | 6 | 1
  End of Re-treatment, Cycle 2, Satisfied | 6 | 1

14. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): Fatigue, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: mITT population was the primary efficacy population and corresponded to all randomized subjects who has a baseline PGA and at least one postbaseline PGA.
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 44 | 43
  Prior to Re-treatment, Cycle 1, Satisfied | 13 | 7
  End of Re-treatment, Cycle 1, Satisfied | 20 | 6
  Prior to Re-treatment, Cycle 2, Satisfied | 7 | 2
  End of Re-treatment, Cycle 2, Satisfied | 9 | 2

15. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): How Others Respond to Your Personal Appearance at Work/School, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: mITT) population was the primary efficacy population and corresponded to all randomized subjects who had a baseline PGA and at least one postbaseline PGA.
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 50 | 48
  Prior to Re-treatment, Cycle 1, Satisfied | 20 | 7
  End of Re-treatment, Cycle 1, Satisfied | 28 | 9
  Prior to Re-treatment, Cycle 2, Satisfied | 7 | 2
  End of Re-treatment, Cycle 2, Satisfied | 8 | 1

16. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): How Your Skin Affects Your Social and Leisure Activities, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 56 | 45
  Prior to Re-treatment, Cycle 1, Satisfied | 23 | 9
  End of Re-treatment, Cycle 1, Satisfied | 29 | 8
  Prior to Re-treatment, Cycle 2, Satisfied | 8 | 0
  End of Re-treatment, Cycle 2, Satisfied | 9 | 0

17. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): How Satisfied Were You With Your Psoriasis Treatment in General? at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 14
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 84 | 79
  Prior to Re-treatment, Cycle 1, Satisfied | 30 | 13
  End of Re-treatment, Cycle 1, Satisfied | 39 | 17
  Prior to Re-treatment, Cycle 2, Satisfied | 7 | 4
  End of Re-treatment, Cycle 2, Satisfied | 10 | 4

18. Secondary Outcome: Patient Psoriasis Satisfaction Questionnaire (PSSQ): I Would Like to Continue With my Current Psoriasis Treatment, at Baseline, Before Retreatment, and at the End of Retreatment
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: as for outcome 14
Measure: Number; unit: Number of Participants
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Number of Participants
  Baseline, Subjects Satisfied | 82 | 78
  Prior to Re-treatment, Cycle 1, Satisfied | 34 | 16
  End of Re-treatment, Cycle 1, Satisfied | 41 | 18
  Prior to Re-treatment, Cycle 2, Satisfied | 11 | 4
  End of Re-treatment, Cycle 2, Satisfied | 10 | 4

19. Secondary Outcome: Physician Global Assessment (PGA) of Disease Activity at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: The modified intent-to-treat (mITT) population will be the primary efficacy population and will correspond to all randomized subjects who have a baseline PGA and at least one postbaseline PGA.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Stop Arm | Maintenance Arm
Number analyzed (Participants) | 86 | 84
Units on a scale | 1.8 (1.02) | 1.4 (1.00)

ADVERSE EVENTS:
Time Frame: Post baseline period
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Stop Arm | Maintenance Arm
Serious Adverse Events (participants affected / at risk) | 6/87 | 4/84
Other Adverse Events (participants affected / at risk) | 25/87 | 32/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stop Arm (N=87) | Maintenance Arm (N=84)
Angina Pectoris (Cardiac disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Bacterial Pyelonephritis (Infections and infestations) | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1
Viith Nerve Paralysis (Gastrointestinal disorders) | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial Stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stop Arm (N=87) | Maintenance Arm (N=84)
Bronchitis (Infections and infestations) | 5 | 9
Nasopharyngitis (Infections and infestations) | 10 | 22
Pharyngitis (Infections and infestations) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 6

LIMITATIONS AND CAVEATS:
Enrollment in this study was slower than expected. Thus, recruitment was terminated early and only 58 percent of planned participants were randomized. As a result, no hypothesis testing was conducted and only descriptive statistics are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.